CLINICAL TRIAL: NCT00086450
Title: Future Revascularization Evaluation in Patients With Diabetes Mellitus: Optimal Management of Multivessel Disease (FREEDOM)
Brief Title: Comparison of Two Treatments for Multivessel Coronary Artery Disease in Individuals With Diabetes (FREEDOM)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Valentin Fuster (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Valentin Fuster, Physician-in-Chief, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCO 02-0163; U01HL071988 (NIH); R01 HL71988
Record Dates: First submitted 2004-07-01; First posted 2004-07-05 (Estimated); Results first posted 2017-02-06 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2016-12

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Diabetes Mellitus; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Diabetes Mellitus; Heart Diseases | interventions — Coronary Artery Bypass; Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Coronary Artery Bypass Graft (Active Comparator): Coronary Artery Bypass Graft
  Interventions: Procedure: Coronary Artery Bypass Graft
- Percutaneous Coronary Intervention (Experimental): Percutaneous Coronary Intervention
  Interventions: Device: Percutaneous Coronary Intervention

INTERVENTIONS:
Procedure: Coronary Artery Bypass Graft — For CABG, participants will receive general anesthesia and will have a breathing tube placed in their throat and they will be unconscious during the operation. An incision is made through the chest bone and muscle, which allows the surgeon access to the heart and diseased vessels. The surgeon will use one or more healthy vessels (either from an artery in the shoulder or a vein in the leg) and will bypass the diseased vessel with the healthy vessel(s). This bypass will provide needed blood supply to the heart.
  Other Names: CABG
  Arms: Coronary Artery Bypass Graft
Device: Percutaneous Coronary Intervention — For PCI, the participant will have two or more drug-eluting stents permanently implanted in their clogged arteries. Drug-eluting stents are coated with a drug that may prevent the disease in the vessel from coming back. The brand names of the stents used in this study are TAXUS and CYPHER.
  The participant will receive a local anesthetic. A small puncture will be made and a balloon-tipped catheter is introduced through the small puncture in the leg/arm and advanced through the artery to the diseased heart vessel. The balloon is then inflated to enlarge the opening in the vessel. After enlarging the vessel, the drug-eluting stent will be placed using a similar balloon catheter. This balloon will be inflated, expanding the stent and placing it in the diseased vessel. Once the stent is fully expanded, the balloon is deflated and removed, leaving the stent in place in the artery.
  Other Names: PCI
  Arms: Percutaneous Coronary Intervention

SUMMARY:
The purpose of this study is to compare 5-year mortality rates in diabetic individuals with multivessel coronary artery disease (CAD) who undergo either coronary artery bypass grafting (CABG) surgery or percutaneous coronary stenting.

DETAILED DESCRIPTION:
BACKGROUND:

The study addresses the critically important problem of how to best revascularize diabetic individuals with multivessel CAD. CAD and diabetes diagnoses are increasing at alarming rates, and much of the information regarding optimal revascularization comes from the Bypass Angioplasty Revascularization Investigation (BARI) study. After five years, data from the BARI study showed 15 excess deaths for every 100 diabetic participants revascularized by percutaneous coronary intervention (PCI) compared to CABG, and at 7 years there were more than 20 deaths. These findings provide compelling evidence for some physicians to conclude that diabetic patients with multivessel disease in need of revascularization are best handled by CABG. But a consensus has not yet been reached because these findings have not been uniformly confirmed by registries and other studies. With the recent introduction of coated stents that significantly reduce or eliminate restenosis, a prevailing belief is that adequate revascularization can be achieved by PCI even in diabetic individuals. New developments in percutaneous techniques should translate to improved prognosis to offset the advantage of CABG seen in the BARI study. Since these new drug eluting stents are not yet approved and are not likely to be on the market for several years, a small window of time exists to gather the evidence to support the strategy that provides optimal revascularization in diabetic individuals.

DESIGN NARRATIVE:

FREEDOM (Future Revascularization Evaluation in Patients with Diabetes Mellitus: Optimal Management of Multivessel Disease) is a multicenter, two-arm, open label, prospective, randomized superiority trial with equal allocation, of 5 years duration with a minimum of 3 years of follow-up. The main objective of the study is to evaluate whether PCI with drug-eluting stenting (PCI/DES) is more or less effective than the existing standard of care, CABG. The study population will consist of 2,400 adults with diabetes mellitus (Type 1 or Type 2) with angiographically confirmed multivessel CAD and morphology amenable to either PCI or CABG, with indication for revascularization based upon symptoms or angina and/or objective evidence of myocardial ischemia. Patients who consent will be randomized on a 1:1 basis either to CABG or multivessel stenting using drug-eluting stents, and followed at 30 days, 1 year, and then annually for at least 3 years, but up to 5 years. A registry of 2000 patients will also be recruited concurrently, comprised of eligible non-consenting patients for the randomized trial. Eligible patients will be randomized to receive either CABG or multivessel stenting using drug-eluting stents. Patients randomized to the PCI/DES arm will receive, at the discretion of the primary physician or interventionalists, either CYPHER Sirolimus eluting stent (Cordis Corporation, Warren, NJ, USA) or the TAXUS paclitaxel-eluting stent (Boston Scientific Corporation, Natick, MA, USA). However, it is intended that only one type of drug-eluting stent be used in a given patient during the course of the trial. The primary outcome of the study is the composite of all-cause mortality, nonfatal myocardial infarction, and stroke at the end of the 5-year patient accrual and follow-up period (minimum follow-up is 3 years). The main secondary endpoint that will be assessed is the 1-year major adverse cardiac and cerebrovascular event (MACCE) rates, including the first of one of the following: death, myocardial infarction, stroke, or repeat revascularization. Additional secondary endpoints include: all-cause and cardiovascular mortality at 1, 2, and 3 years; rates of individual MACCE endpoints at 30 days post-procedure; quality of life at 30 days, 6 months, and annually post-procedure; long term costs and cost-effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus (Type 1 or Type 2), defined according to the American Diabetes Association as either:

  1. presence of classic symptoms of diabetes mellitus with unequivocal elevation of plasma glucose (2-hour post-prandial or random of greater than 200 mg/dL (11mmol/L) or
  2. fasting plasma glucose elevation on more than one occasion of at least 126 mg/dL (7mmol/L)
* Currently undergoing pharmacological or non-pharmacological treatment for diabetes
* Angiographically confirmed multivessel CAD [critical (greater than or equal to 70%) lesions in at least two major epicardial vessels and in at least two separate coronary artery territories (LAD, LCX, RCA)] amenable to either PCI or CABG
* Angiographic characteristics amendable to both PCI/DES and CABG
* Indication for revascularization based upon symptoms of angina and/or objective evidence of myocardial ischemia

Exclusion Criteria:

* Severe congestive heart failure (class III or IV according to New York Heart Association [NYHA] or pulmonary edema)
* Prior CABG surgery
* Prior valve surgery
* Prior PCI with stent implantation within 6 months of study entry
* Stroke within 6 months of study entry; if stroke occurred more than 6 months prior to study entry, must have significant residual neurologic involvement, as reflected in a Rankin Score of greater than 1
* Prior history of significant bleeding (within 6 months of study entry) that may occur during CABG or PCI/DES related anticoagulation
* In-stent restenosis of a target vessel
* Two or more chronic total occlusions in major coronary territories
* Left main stenosis (at least 50% diameter stenosis)
* Acute ST-elevation MI (Q-wave) within 72 hours of study entry requiring revascularization
* Abnormal creatine kinase level (greater than twice the normal limit); or abnormal CK-MB level at study entry
* Planned simultaneous surgical procedure unrelated to coronary revascularization (e.g., valve repair/replacement, aneurysmectomy, carotid endarterectomy, or carotid stent)
* Cannot undergo either CABG or PCI/DES because of a coexisting medical condition
* Significant leukopenia, neutropenia, thrombocytopenia, anemia, or known bleeding diathesis
* Intolerance to aspirin or both clopidogrel and ticlopidine
* Dementia with a score of less than 20 on the Mini Mental Status Examination (MMSE)
* Extra-cardiac illness that is expected to limit survival to less than 5 years (e.g., oxygen-dependent chronic obstructive pulmonary disease, active hepatitis, significant hepatic failure, or severe kidney disease)
* Pregnant
* Currently enrolled in another clinical trial
* Unable to attend required follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1900 (Actual)
Dates: Start 2004-04; Primary Completion 2012-07 (Actual); Study Completion 2018-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Valentin Fuster, Study Chair — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Derived] Takahashi K, Serruys PW, Fuster V, Farkouh ME, Spertus JA, Cohen DJ, Park SJ, Park DW, Ahn JM, Onuma Y, Kent DM, Steyerberg EW, van Klaveren D; SYNTAX, BEST, and FREEDOM Trial investigators. External Validation of the FREEDOM Score for Individualized Decision Making Between CABG and PCI. J Am Coll Cardiol. 2022 Apr 19;79(15):1458-1473. doi: 10.1016/j.jacc.2022.01.049. PMID 35422242
- [Derived] Esper RB, Farkouh ME, Ribeiro EE, Hueb W, Domanski M, Hamza TH, Siami FS, Godoy LC, Mathew V, French J, Fuster V. SYNTAX Score in Patients With Diabetes Undergoing Coronary Revascularization in the FREEDOM Trial. J Am Coll Cardiol. 2018 Dec 11;72(23 Pt A):2826-2837. doi: 10.1016/j.jacc.2018.09.046. PMID 30522646
- [Derived] Farkouh ME, Domanski M, Dangas GD, Godoy LC, Mack MJ, Siami FS, Hamza TH, Shah B, Stefanini GG, Sidhu MS, Tanguay JF, Ramanathan K, Sharma SK, French J, Hueb W, Cohen DJ, Fuster V; FREEDOM Follow-On Study Investigators. Long-Term Survival Following Multivessel Revascularization in Patients With Diabetes: The FREEDOM Follow-On Study. J Am Coll Cardiol. 2019 Feb 19;73(6):629-638. doi: 10.1016/j.jacc.2018.11.001. Epub 2018 Nov 11. PMID 30428398
- [Derived] van Diepen S, Fuster V, Verma S, Hamza TH, Siami FS, Goodman SG, Farkouh ME. Dual Antiplatelet Therapy Versus Aspirin Monotherapy in Diabetics With Multivessel Disease Undergoing CABG: FREEDOM Insights. J Am Coll Cardiol. 2017 Jan 17;69(2):119-127. doi: 10.1016/j.jacc.2016.10.043. PMID 28081820
- [Derived] Dangas GD, Farkouh ME, Sleeper LA, Yang M, Schoos MM, Macaya C, Abizaid A, Buller CE, Devlin G, Rodriguez AE, Lansky AJ, Siami FS, Domanski M, Fuster V; FREEDOM Investigators. Long-term outcome of PCI versus CABG in insulin and non-insulin-treated diabetic patients: results from the FREEDOM trial. J Am Coll Cardiol. 2014 Sep 23;64(12):1189-97. doi: 10.1016/j.jacc.2014.06.1182. PMID 25236509
- [Derived] Abdallah MS, Wang K, Magnuson EA, Spertus JA, Farkouh ME, Fuster V, Cohen DJ; FREEDOM Trial Investigators. Quality of life after PCI vs CABG among patients with diabetes and multivessel coronary artery disease: a randomized clinical trial. JAMA. 2013 Oct 16;310(15):1581-90. doi: 10.1001/jama.2013.279208. PMID 24129463
- [Derived] Farkouh ME, Boden WE, Bittner V, Muratov V, Hartigan P, Ogdie M, Bertolet M, Mathewkutty S, Teo K, Maron DJ, Sethi SS, Domanski M, Frye RL, Fuster V. Risk factor control for coronary artery disease secondary prevention in large randomized trials. J Am Coll Cardiol. 2013 Apr 16;61(15):1607-15. doi: 10.1016/j.jacc.2013.01.044. PMID 23500281
- [Derived] Magnuson EA, Farkouh ME, Fuster V, Wang K, Vilain K, Li H, Appelwick J, Muratov V, Sleeper LA, Boineau R, Abdallah M, Cohen DJ; FREEDOM Trial Investigators. Cost-effectiveness of percutaneous coronary intervention with drug eluting stents versus bypass surgery for patients with diabetes mellitus and multivessel coronary artery disease: results from the FREEDOM trial. Circulation. 2013 Feb 19;127(7):820-31. doi: 10.1161/CIRCULATIONAHA.112.147488. Epub 2012 Dec 31. PMID 23277307
- [Derived] Farkouh ME, Domanski M, Sleeper LA, Siami FS, Dangas G, Mack M, Yang M, Cohen DJ, Rosenberg Y, Solomon SD, Desai AS, Gersh BJ, Magnuson EA, Lansky A, Boineau R, Weinberger J, Ramanathan K, Sousa JE, Rankin J, Bhargava B, Buse J, Hueb W, Smith CR, Muratov V, Bansilal S, King S 3rd, Bertrand M, Fuster V; FREEDOM Trial Investigators. Strategies for multivessel revascularization in patients with diabetes. N Engl J Med. 2012 Dec 20;367(25):2375-84. doi: 10.1056/NEJMoa1211585. Epub 2012 Nov 4. PMID 23121323
- [Derived] Bansilal S, Farkouh ME, Hueb W, Ogdie M, Dangas G, Lansky AJ, Cohen DJ, Magnuson EA, Ramanathan K, Tanguay JF, Muratov V, Sleeper LA, Domanski M, Bertrand ME, Fuster V. The Future REvascularization Evaluation in patients with Diabetes mellitus: optimal management of Multivessel disease (FREEDOM) trial: clinical and angiographic profile at study entry. Am Heart J. 2012 Oct;164(4):591-9. doi: 10.1016/j.ahj.2012.06.012. PMID 23067919

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All trial-eligible patients must have multivessel disease suitable for either approach as determined by both an interventional cardiologist and a surgical investigator. The interventionalist and surgeon at each site will document their intentions of which vessels are targets for revascularization.
Period: Overall Study
Arm/Group | Percutaneous Coronary Intervention | Coronary Artery Bypass Graft
Started | 953 | 947
Completed | 953 | 947
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Percutaneous Coronary Intervention | Coronary Artery Bypass Graft | Total
Number analyzed (Participants) | 953 | 947 | 1900
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (8.9) | 63.1 (9.2) | 63.1 (9.1)
Gender [Count of Participants; unit: Participants]
  Female | 255 | 289 | 544
  Male | 698 | 658 | 1356

OUTCOME MEASURES:

1. Primary Outcome: 5-year Composite Endpoint of All-cause Mortality, Non-fatal Myocardial Infarction, and Stroke
Description: median 3.8 years of follow-up
Time Frame: Measured at Year 5
Measure: Number; unit: percentage of participants
Arm/Group | Percutaneous Coronary Intervention | Coronary Artery Bypass Graft
Number analyzed (Participants) | 953 | 947
percentage of participants | 26.6 | 18.7
Statistical Analysis 1: Comparison: Percutaneous Coronary Intervention vs Coronary Artery Bypass Graft; Test type: Superiority or Other; p = 0.005, Regression, Cox; Cox Proportional Hazard = 7.9, 95% CI [3.3 to 12.5]

2. Secondary Outcome: Major MACCE Rates, Including the First of One of the Following: Death, Myocardial Infarction, Stroke, or Repeat Revascularization
Time Frame: Measured at Year 1
Measure: Number; unit: percentage of participants
Arm/Group | Percutaneous Coronary Intervention | Coronary Artery Bypass Graft
Number analyzed (Participants) | 953 | 947
percentage of participants | 16.8 | 11.8
Statistical Analysis 1: Comparison: Percutaneous Coronary Intervention vs Coronary Artery Bypass Graft; Test type: Superiority or Other; p = 0.004, Regression, Cox; Hazard Ratio (HR) = 2.74, 95% CI [1.91 to 3.89]

3. Secondary Outcome: All-cause Mortality
Time Frame: Measured at Year 5
Measure: Number; unit: percentage of participants
Arm/Group | Percutaneous Coronary Intervention | Coronary Artery Bypass Graft
Number analyzed (Participants) | 953 | 947
percentage of participants | 16.3 | 10.9
Statistical Analysis 1: Comparison: Percutaneous Coronary Intervention vs Coronary Artery Bypass Graft; Test type: Superiority or Other; p = 0.049, Log Rank; Hazard Ratio (HR) = 5.4

4. Secondary Outcome: Rates of Individual MACCE Endpoints
Description: Major adverse cardiovascular and cerebrovascular events
Time Frame: Measured at Day 30
Measure: Number; unit: percentage of participants
Arm/Group | Percutaneous Coronary Intervention | Coronary Artery Bypass Graft
Number analyzed (Participants) | 953 | 947
percentage of participants | 4.8 | 5.2
Statistical Analysis 1: Comparison: Percutaneous Coronary Intervention vs Coronary Artery Bypass Graft; Test type: Superiority or Other; p = 0.68, Regression, Cox

ADVERSE EVENTS:
Arm/Group | Percutaneous Coronary Intervention | Coronary Artery Bypass Graft
Serious Adverse Events (participants affected / at risk) | 24/953 | 42/947
Other Adverse Events (participants affected / at risk) | 44/953 | 37/947
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Percutaneous Coronary Intervention (N=953) | Coronary Artery Bypass Graft (N=947)
Major bleeding (Blood and lymphatic system disorders) | 23 (23) | 34 (34)
Acute Renal Failure (Renal and urinary disorders) | 1 (1) | 8 (8)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Percutaneous Coronary Intervention (N=953) | Coronary Artery Bypass Graft (N=947)
Renal insufficiency (Renal and urinary disorders) | 44 (44) | 37 (37)

LIMITATIONS AND CAVEATS:
Since the trial was not blinded, patients may have been treated differently on the basis of their surgical procedure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes